CLINICAL TRIAL: NCT01349595
Title: Impact of Proteasome Inhibition on Anti-Donor HLA Antibody Production After Kidney Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted due to lack of funding
Sponsor: Mark Stegall (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark Stegall, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-001487
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Disorder of Transplanted Kidney
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bortezomib (Experimental): Bortezomib is a type of targeted chemotherapy
  Interventions: Drug: Bortezomib
- Standard Post-transplant Treatment (No Intervention): Mayo Clinic standard post kidney transplant follow-up.

INTERVENTIONS:
Drug: Bortezomib — Patients randomized to bortezomib treatment will receive 2, 4-dose cycles of drug followed by a 2 month "hiatus". At the end of this time, subjects will be re-evaluated for the appropriateness of receiving a 3rd and 4th cycle of bortezomib. Bortezomib will be given subcutaneously (under the skin). If unable to give subcutaneously, bortezomib will be given as a single IV (injection into vein) over a time of 3 to 5 seconds. Patients will receive up to 4, four-dose cycles of 1.3 mg/m(2) (based on body surface area).
  Other Names: Velcade
  Arms: Bortezomib

SUMMARY:
The purpose of this study is to see if treating patients who have high levels of donor specific alloantibodies post-transplant with bortezomib might prevent the development of transplant glomerulopathy and preserve allograft function.

ELIGIBILITY:
Inclusion Criteria:

* Female subject is either postmenopausal for at least 1 year before the screening visit, surgically sterilized, or if they are of childbearing potential agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse.
* Male subjects, even if surgically sterilized (i.e. status postvasectomy), must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug or completely abstain from heterosexual intercourse.
* Kidney transplant recipients (living and deceased donors) who received a transplant in the last 3 years and have high Donor Specific Antibody (DSA) levels (defined as Mean Fluorescent Intensity levels >2000 by solid phase and single antigen bead LABscreen assays).

Exclusion Criteria:

* Patients who are recipients of ABO (blood type) incompatible kidney transplants.
* Patient with an Glomerular Filtration Rate (eGFR) ≤30 m/min at time of study entry.
* Patient with biopsy proven transplant glomerulopathy (Banff 2007 - cg score ≥2) within 2 months prior to randomization.
* Patients with biopsy-proven acute rejection at the time of randomization defined as Acute Cellular Rejection Patients with documented biopsy proven recurrence of disease or de novo glomerular disease post-transplant prior to enrollment.
* Patient has a platelet count of <30 x 10(9)/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of <1.0 x 10(9)/L within 14 days before enrollment.
* Patient has a history of post-transplant neutropenia on mycophenolate based immunosuppressive therapy.
* Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >3 times upper limit of normal [ULN]) at screening.
* Patient has >1.5 x ULN Total Bilirubin.
* Patient had any history of myocardial infarction in the past 3 years prior to enrollment or has New York Heart Association (NYHA) Class II to IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron, or mannitol.
* Female subject is pregnant or lactating.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Cytomegalovirus (CMV) sero-negative recipients who received a transplant from a CMV-sero-positive donor.(CMV- recipients of CMV- donor kidneys are acceptable)
* Epstein Barr Virus (EBV) sero-negative recipients.
* History of CMV + or EBV + viremia since transplantation.
* History of SPELL OUT HCV positivity (by PCR).
* History of Post-transplant lymphoproliferative disease.
* History of polyoma virus nephropathy or BK virus viremia (peripheral blood viral load of 5000 to 5,000,000 copies/mL).
* Patients who are HIV-positive or HBsAg-positive.
* Recipients of a kidney from a donor who tests positive for HIV, HBsAg or anti-HCV.
* Patients with current or recent severe systemic (pathogen detected in blood or Cerebrospinal fluid) infections within the 4 weeks prior to randomization.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patient is currently receiving everolimus, sirolimus, or azathioprine as one of the immunosuppressive agents and intends to remain on this regimen.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Inability to perform followup or to undergo protocol biopsy.
* Active diabetic neuropathy at the time of treatment initiation.
* Patient has ≥Grade 2 peripheral neuropathy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic transplant program in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Bortezomib | Standard Post-transplant Treatment
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Lack of funding | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib | Standard Post-transplant Treatment | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of a Combined Endpoint of Death-censored Graft Loss or Greater Than 50% Reduction in Estimated Glomerular Filtration (eGFR) in Study Subjects.
Time Frame: 60 months after enrollment in the study
Population: Results data for zero participants were analyzed; long-term follow-up evaluation of participants was not possible due to discontinuation of funding.
Arm/Group | Bortezomib | Standard Post-transplant Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 months after kidney transplantation
Arm/Group | Bortezomib | Standard Post-transplant Treatment
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=2) | Standard Post-transplant Treatment (N=2)
nausea/vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) — Evening of drug infusions
fatigue (General disorders) | 2 (2) | 0 (0)
Pain at injection site (General disorders) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) — Bilateral shooting pain down side of legs x 30 minutes

LIMITATIONS AND CAVEATS:
Although subjects completed the cycles of drug, long term follow-up visits were not possible due to funding discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes